CLINICAL TRIAL: NCT04250857
Title: HeartStart FRx Defibrillator Event Registry
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: MATC-ECR-Registry-2018-10295
Record Dates: First submitted 2019-12-18; First posted 2020-01-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Suspected Sudden Cardiac Arrest: All subject with suspected of a circulatory arrest for any cause.
  Interventions: Device: HeartStart FRX

INTERVENTIONS:
Device: HeartStart FRX — Automated External Defibrillator

SUMMARY:
This post market clinical follow-up study is a multi-center, non-randomized, unblinded, observational registry of the performance of the FRx Automated external defibrillator (AED) used in conjunction with electrodes with or without use of the infant/child key. The registry is focused only on on post-event data collection and does not prescribe any device usage. This registry has several safeguards in place to prevent against selections bias, including enrollment of all participants who have pads placed. This registry will evaluate the safety and verify the clinical performance of the device in relation to its claims, when used in accordance with the Device Manual.

ELIGIBILITY:
Inclusion Criteria:

* Subjects accepted into the study must: have been suspected of a circulatory arrest for any cause
* Have had HeartStart FRx AED with electrodes: HeartStart SMART PADS II applied to their body and powered up, regardless of whether a defibrillation shock was delivered

Exclusion Criteria:

* AED or pad use other than the HeartStart FRx AED with electrodes : HeartStart SMART PADS II
* AED used for training purposes.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Use of the HeartStart FRx AED is intended for the following populations in addition to adults: newborns, neonates, infant, children, and adolescents. It may also be used on pregnant women. Devices are located in public access spaces and with first responders around the world.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Algorithm accuracy | Up to 15 minutes after device placement
  Algorithm performance as determined by adjudication of the wave form data as aligned with the device advisement.
Shock Delivery | 1 day
  Percentage of events where a shock was delivered when indicated.
Unexpected adverse events. | 1 day
  Frequency and severity of unexpected adverse events.
Unanticipated adverse device effects (UADE) | 1 day
  Unanticipated adverse device effects (UADE)

SECONDARY OUTCOMES:
Time Intervals | 1 day
  Measurements of device performance time intervals.
Device Preparation | 1 day
  Percentage of events where the device prepared to shock.
Shock Energy Delivered | 1 day
  The amount of shock energy delivered as measured in joules with each shock.
Pad Replacement | 1 day
  Frequency of pad replacement.
User | 1 day
  Frequency of user pressing the shock button.

CONTACTS AND LOCATIONS:
Locations (1):
- Philips, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No